CLINICAL TRIAL: NCT05610462
Title: A Multicenter Randomized Controlled Trial of Exercise in Aortic Dissection Survivors
Brief Title: Trial of Exercise in Aortic Dissection Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Washington University School of Medicine (Other); University of Michigan (Other); John Ritter Foundation for Aortic Health (Unknown)
Responsible Party: Principal Investigator, Siddharth Prakash, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-22-0936
Record Dates: First submitted 2022-10-27; First posted 2022-11-09 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Thoracic Aortic Dissection
Keywords: Thoracic Aortic Disease; Ambulatory Blood Pressure; Arterial stiffness; Aortic Dissection; Mental Health; Exercise
MeSH Terms: conditions — Dissection, Thoracic Aorta; Aortic Dissection; Psychological Well-Being; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Control (Active Comparator): Participants who are randomized to usual care will attend routine clinic visits but will not receive any teaching or supervision and will not participate in any in-person or virtual exercise sessions. Instead, they will receive standardized counseling about exercise, including an exercise pamphlet that is given to all thoracic aortic dissection (TAD) patients.
  Interventions: Behavioral: Usual Care
- Guided Exercise Training Program (Experimental): Participants who are randomized to the guided exercise group will undergo initial training that consists of: one video demonstration, one exercise training session or group session, one follow up home visit, and virtual check-ins.
  Interventions: Behavioral: Guided Exercise Training Program

INTERVENTIONS:
Behavioral: Guided Exercise Training Program — The guided exercise program training consists of: a video demonstration, an exercise training session or group session, a follow up home visit, and virtual check-ins. The exercises include treadmill, wall sits, straight leg raise, bicep curls, hand grips with dynamometer at 40% maximal voluntary contraction (MVC), and Stationary cycling at moderate intensity (100 Watts).
  Arms: Guided Exercise Training Program
Behavioral: Usual Care — Usual care consists of routine clinic visits and standardized counseling about exercise, including an exercise pamphlet that is given to all thoracic aortic dissection (TAD) patients.
  Arms: Usual Care Control

SUMMARY:
The primary objective of this study is to test the safety and mental health benefits of a guided exercise program for people who survived an acute aortic dissection. This study is designed to answer several questions:

1. Can supervised exercise improve confidence and mental health in dissection survivors?;
2. How safe are different types of exercise for people who are living with severe aortic disease?;
3. Can tests be developed to determine rational and safe limits to guide exercise recommendations for individual patients?;
4. Does the blood pressure response to exercise predict risks for aortic enlargement or dissection in unique ways that other tests may not detect?

The long-term goal of this research is to develop new guidelines for exercise and daily activities that promote the safety and well-being of all TAD patients.

All participants will be required to:

* Complete online questionnaires (demographic survey, 2009 Behavioral Risk Factor Surveillance Survey, the Patient-Reported Outcomes Measurement Information System 29 (PROMIS-29) v2.0 profile questionnaire)
* Exercise (>150 minutes/week)
* Receive all usual clinically indicated care, including diagnostic tests and medications. Recommendations for tests or interventions will not change based on the assigned study arm.

Participants who are randomized to guided exercise group will undergo initial training that consists of: one video demonstration, one exercise training session or group session, one follow up home visit, and virtual check-ins.

Participants who are randomized to usual care will attend routine clinic visits but will not receive any teaching or supervision and will not participate in any in-person or virtual exercise sessions. Instead, they will receive standardized counseling about exercise, including an exercise pamphlet that is given to all TAD patients.

DETAILED DESCRIPTION:
Required number of study visits: 6 (3 in-person, 3 virtual)

Estimated total visit time per participant: 8 hours (guided exercise arm), 4 hours (control arm)

* Visit 1 (Enrollment): After confirmation of eligibility and consent, participants will complete a demographic survey (age, sex, race, ethnicity) and the PROMIS-29 v2.0 profile questionnaire, which is validated to assess seven health domains (physical function, fatigue, pain, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance). Arterial pressure waveform and pulse wave velocity analysis will be performed (Sphygmocor, AtCor Medical, Inc.) and one set of orthostatic vital signs will be recorded (sitting x 3, lying, standing). Consent will also be obtained to extract additional outcome data from health records.
* Visit 2 (Supervised training session): Participants will be fitted with ambulatory blood pressure monitors (ABPM, OnTrak, Space Labs, Inc.) and will complete an exercise circuit under the supervision of basic life support (BLS)-certified personnel. Participants will maintain each exercise at target intensity for at least 1 minute, or long enough to record at least one measurement. At steady state exertion, spotters will manually trigger OnTrak readings. Participants will pause between each exercise long enough to complete one ABPM reading (3 minutes). The circuit will be repeated once so that there will be two sets of measurements per exercise. Participants will rate their perceived level of exertion on a modified Borg scale.
* In all cases, a spotter will brace the arm during ABPM measurements and ensure that pressures are recorded: Modified treadmill, wall sits, straight leg raises, bicep curls, hand grips with dynamometer at 40% maximum voluntary contraction (MVC) on the dominant arm.

Participants will then receive individualized instruction about how to implement this exercise protocol at home. The study team will promote a weekly target 5 days or at least 150 total minutes of exercise. Participants will complete a survey about where they intend to exercise (in their home or in a gym) and the type of equipment that they plan to use (a treadmill, a bicycle, or both). They will also be counseled to record their activities in an exercise diary. If they have a home blood pressure cuff or wearable device that can record fitness data, they will send the digital files to the study team at UTHealth. The instructional video and a diary template document will be emailed to all participants.

* Visit 3 (Long Virtual Check-in): In the first month after enrollment, the study teams will conduct one video check-in with each participant to assess their home exercise setup, reinforce teaching about the exercise circuit, and answer questions about exercise. During the check-in, they will also observe and correct participants while they perform each exercise.
* Visits 4 and 5 (Short Virtual Check-ins): Shorter video visits without exercise demonstrations will be repeated at 3 and 9 months after enrollment. These visits will be conducted in group sessions where participants will be encouraged to share their experiences with the exercise protocol and to troubleshoot potential obstacles to exercise. Participants will also transmit home blood pressure or fitness data to UTHealth if they are available. The study teams will promote the target of more than 150 minutes of moderate exercises per week at each interaction. All participants will also receive digital REDCap surveys about the intensity and frequency of their activities at 1, 3, and 9 months, and at the conclusion of the study. The content will be the same as the initial survey with an additional link to send messages directly to the study team.
* Visit 6 (End of study visit): All study participants will undergo office blood pressure and Sphygmocor measurements and complete the same BRFSS activity and PROMIS-29 v2.0 questionnaires as at enrollment. They will be asked to wear an ABPM for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

-Patients who survived a thoracic aortic dissection (Type A or B) at least 3 months prior to study.

Exclusion Criteria:

* Routine participation in > 150 minutes per week of moderate intensity exercises
* Unable to attend at least one exercise training session in person
* Uncontrolled hypertension: mean SBP > 160 mmHg at rest
* Symptomatic aortic, coronary, or vascular disease
* Unable to complete exercise circuit due to physical limitations, equipment, space, or time commitment
* Do not own a treadmill or stationary cycle or have regular access to one at a gym.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-01-28 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with clinically important difference (CID) in the PROMIS-29 T score or the PROMIS mental health summary score | Change from baseline PROMIS-29 T score at 12 months
  The primary outcome is a clinically significant change in the PROMIS-29 T score or the PROMIS mental health summary score, a subset of PROMIS questions that primarily assess emotional distress (anxiety and depressive symptoms). The minimum clinically important difference (CID) is 5 points.

SECONDARY OUTCOMES:
Change in office blood pressure | Change in office systolic and diastolic blood pressure at 12 months
  The mean of three seated brachial measurements will be measured in the non-dominant arm.
Change in daytime ambulatory hypertensive burden | Change in systolic and diastolic hypertensive burden by ABPM at 12 months
  In 24 hour ambulatory blood pressures, the % of daytime systolic readings > 135 or diastolic readings > 80 mmHg
Change in nighttime ambulatory hypertensive burden | Change in systolic and diastolic hypertensive burden by ABPM at 12 months
  In 24 hour ambulatory blood pressures, the % of nighttime systolic readings > 120 or diastolic readings > 65 mmHg
Prevalence of exertional hypertension | 1 month, at study visit 2
  Any systolic pressure > 180 mmHg, any diastolic pressure > 110 mmHg, or > 50 mmHg increase in systolic or diastolic pressures with exercise
Change in ambulatory nocturnal dipping | Change in nocturnal dipping by ABPM at 12 months
  In 24 hour ambulatory blood pressure, the % drop in mean nighttime pressures compared to mean daytime pressures.
Change in aortic augmentation index | Change in aortic augmentation index at 12 months
  Aortic augmentation index will be measured using the Sphygmocor XCEL device
Change in pulse wave velocity | Change in pulse wave velocity at 12 months
  Carotid-femoral pulse wave velocity will be measured using the Sphygmocor XCEL device.
Change in exercise minutes | Change in exercise minutes between study enrollment and 3 months, 9 months and 12 months.
  Minutes of moderate or high intensity exercise per week, as self-assessed by patients on BRFSS questionnaires
Change in grip strength | Change in grip strength at 12 months
  Maximum grip strength as measured by dynamometer in Kg
Change in antihypertensive medications | Change in antihypertensive medications at 12 months
  Number of antihypertensive medications x total dosage in mg
Total study time as a proportion of clinical time | 12 months
  Logged time of all study-specific encounters divided by the estimated total time spent in clinically indicated interactions for TAD surveillance or treatment, ascertained from medical records
Change in systolic blood pressure with exercise | From baseline to end of study visit (12 months after baseline)
Change in diastolic blood pressure with exercise | From baseline to end of study visit (12 months after baseline)
Post-guided exercise program heart rate | Baseline
Systolic blood pressure recovery times | Baseline
  This is the time taken for the post work out blood pressure to get back to at least 10 percent of baseline blood pressure at enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Siddharth Prakash, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (3):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - University of Texas Health Science Center, Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Januzzi JL, Isselbacher EM, Fattori R, Cooper JV, Smith DE, Fang J, Eagle KA, Mehta RH, Nienaber CA, Pape LA; International Registry of Aortic Dissection (IRAD). Characterizing the young patient with aortic dissection: results from the International Registry of Aortic Dissection (IRAD). J Am Coll Cardiol. 2004 Feb 18;43(4):665-9. doi: 10.1016/j.jacc.2003.08.054. PMID 14975480
- [Background] Chaddha A, Eagle KA, Braverman AC, Kline-Rogers E, Hirsch AT, Brook R, Jackson EA, Woznicki EM, Housholder-Hughes S, Pitler L, Franklin BA. Exercise and Physical Activity for the Post-Aortic Dissection Patient: The Clinician's Conundrum. Clin Cardiol. 2015 Nov;38(11):647-51. doi: 10.1002/clc.22481. PMID 26769698
- [Background] Braverman AC. Medical management of thoracic aortic aneurysm disease. J Thorac Cardiovasc Surg. 2013 Mar;145(3 Suppl):S2-6. doi: 10.1016/j.jtcvs.2012.11.062. Epub 2012 Dec 20. PMID 23260459
- [Background] Milewicz DM, Prakash SK, Ramirez F. Therapeutics Targeting Drivers of Thoracic Aortic Aneurysms and Acute Aortic Dissections: Insights from Predisposing Genes and Mouse Models. Annu Rev Med. 2017 Jan 14;68:51-67. doi: 10.1146/annurev-med-100415-022956. PMID 28099082
- [Background] Milewicz D, Hostetler E, Wallace S, Mellor-Crummey L, Gong L, Pannu H, Guo DC, Regalado E. Precision medical and surgical management for thoracic aortic aneurysms and acute aortic dissections based on the causative mutant gene. J Cardiovasc Surg (Torino). 2016 Apr;57(2):172-7. Epub 2016 Feb 2. PMID 26837258
- [Background] Franz IW, Behr U, Ketelhut R. Resting and exercise blood pressure with atenolol, enalapril and a low-dose combination. J Hypertens Suppl. 1987 Aug;5(3):S37-41. PMID 2822879
- [Background] Virtanen K, Janne J, Frick MH. Response of blood pressure and plasma norepinephrine to propranolol, metoprolol and clonidine during isometric and dynamic exercise in hypertensive patients. Eur J Clin Pharmacol. 1982;21(4):275-9. doi: 10.1007/BF00637613. PMID 7056271
- [Background] Chen X, Hassan MO, Jones JV, Sleight P, Floras JS. Baroreflex sensitivity and the blood pressure response to beta-blockade. J Hum Hypertens. 1999 Mar;13(3):185-90. doi: 10.1038/sj.jhh.1000786. PMID 10204815
- [Background] Hamer M, Bauman A, Bell JA, Stamatakis E. Examining associations between physical activity and cardiovascular mortality using negative control outcomes. Int J Epidemiol. 2019 Aug 1;48(4):1161-1166. doi: 10.1093/ije/dyy272. PMID 30541040
- [Background] Gibson C, Nielsen C, Alex R, Cooper K, Farney M, Gaufin D, Cui JZ, van Breemen C, Broderick TL, Vallejo-Elias J, Esfandiarei M. Mild aerobic exercise blocks elastin fiber fragmentation and aortic dilatation in a mouse model of Marfan syndrome associated aortic aneurysm. J Appl Physiol (1985). 2017 Jul 1;123(1):147-160. doi: 10.1152/japplphysiol.00132.2017. Epub 2017 Apr 6. PMID 28385916
- [Background] Nakayama A, Morita H, Nagayama M, Hoshina K, Uemura Y, Tomoike H, Komuro I. Cardiac Rehabilitation Protects Against the Expansion of Abdominal Aortic Aneurysm. J Am Heart Assoc. 2018 Feb 27;7(5):e007959. doi: 10.1161/JAHA.117.007959. PMID 29487112
- [Background] Bartee S, Shrestha S, Ramos B, Bilbrey T, Carbone P, Schussler JM, Deutsch R, Adams J. Specificity of testing in a cardiac rehabilitation setting resulting in a patient's return to high-intensity outdoor activity following aortic dissection repair. Proc (Bayl Univ Med Cent). 2016 Apr;29(2):151-3. doi: 10.1080/08998280.2016.11929395. PMID 27034550
- [Background] Corone S, Iliou MC, Pierre B, Feige JM, Odjinkem D, Farrokhi T, Bechraoui F, Hardy S, Meurin P; Cardiac Rehabilitation working Group of the French Society of Cardiology. French registry of cases of type I acute aortic dissection admitted to a cardiac rehabilitation center after surgery. Eur J Cardiovasc Prev Rehabil. 2009 Feb;16(1):91-5. doi: 10.1097/HJR.0b013e32831fd6c8. PMID 19237998
- [Background] Ritchey MD, Maresh S, McNeely J, Shaffer T, Jackson SL, Keteyian SJ, Brawner CA, Whooley MA, Chang T, Stolp H, Schieb L, Wright J. Tracking Cardiac Rehabilitation Participation and Completion Among Medicare Beneficiaries to Inform the Efforts of a National Initiative. Circ Cardiovasc Qual Outcomes. 2020 Jan;13(1):e005902. doi: 10.1161/CIRCOUTCOMES.119.005902. Epub 2020 Jan 14. PMID 31931615
- [Background] Robicsek F, Thubrikar MJ. Hemodynamic considerations regarding the mechanism and prevention of aortic dissection. Ann Thorac Surg. 1994 Oct;58(4):1247-53. doi: 10.1016/0003-4975(94)90523-1. PMID 7944800
- [Background] de Virgilio C, Nelson RJ, Milliken J, Snyder R, Chiang F, MacDonald WD, Robertson JM. Ascending aortic dissection in weight lifters with cystic medial degeneration. Ann Thorac Surg. 1990 Apr;49(4):638-42. doi: 10.1016/0003-4975(90)90315-w. PMID 2322060
- [Background] Aparci M, Erdal M, Isilak Z, Yalcin M, Uz O, Arslan Z, Kardesoglu E. Enlargement of the aorta: An occupational disease? Exp Clin Cardiol. 2013 Spring;18(2):93-7. PMID 23940428
- [Background] Finnoff JT, Smith J, Low PA, Dahm DL, Harrington SP. Acute hemodynamic effects of abdominal exercise with and without breath holding. Arch Phys Med Rehabil. 2003 Jul;84(7):1017-22. doi: 10.1016/s0003-9993(03)00049-2. PMID 12881827
- [Background] Chrysant SG. Current evidence on the hemodynamic and blood pressure effects of isometric exercise in normotensive and hypertensive persons. J Clin Hypertens (Greenwich). 2010 Sep;12(9):721-6. doi: 10.1111/j.1751-7176.2010.00328.x. PMID 20883233
- [Background] Salvi P, Grillo A, Marelli S, Gao L, Salvi L, Viecca M, Di Blasio AM, Carretta R, Pini A, Parati G. Aortic dilatation in Marfan syndrome: role of arterial stiffness and fibrillin-1 variants. J Hypertens. 2018 Jan;36(1):77-84. doi: 10.1097/HJH.0000000000001512. PMID 29210860
- [Background] Reddy YNV, Andersen MJ, Obokata M, Koepp KE, Kane GC, Melenovsky V, Olson TP, Borlaug BA. Arterial Stiffening With Exercise in Patients With Heart Failure and Preserved Ejection Fraction. J Am Coll Cardiol. 2017 Jul 11;70(2):136-148. doi: 10.1016/j.jacc.2017.05.029. PMID 28683960
- [Background] Hatzaras IS, Bible JE, Koullias GJ, Tranquilli M, Singh M, Elefteriades JA. Role of exertion or emotion as inciting events for acute aortic dissection. Am J Cardiol. 2007 Nov 1;100(9):1470-2. doi: 10.1016/j.amjcard.2007.06.039. Epub 2007 Aug 22. PMID 17950810
- [Background] Erbel R, Aboyans V, Boileau C, Bossone E, Bartolomeo RD, Eggebrecht H, Evangelista A, Falk V, Frank H, Gaemperli O, Grabenwoger M, Haverich A, Iung B, Manolis AJ, Meijboom F, Nienaber CA, Roffi M, Rousseau H, Sechtem U, Sirnes PA, Allmen RS, Vrints CJ; ESC Committee for Practice Guidelines. 2014 ESC Guidelines on the diagnosis and treatment of aortic diseases: Document covering acute and chronic aortic diseases of the thoracic and abdominal aorta of the adult. The Task Force for the Diagnosis and Treatment of Aortic Diseases of the European Society of Cardiology (ESC). Eur Heart J. 2014 Nov 1;35(41):2873-926. doi: 10.1093/eurheartj/ehu281. Epub 2014 Aug 29. No abstract available. PMID 25173340
- [Background] Chaddha A, Kline-Rogers E, Woznicki EM, Brook R, Housholder-Hughes S, Braverman AC, Pitler L, Hirsch AT, Eagle KA. Cardiology patient page. Activity recommendations for postaortic dissection patients. Circulation. 2014 Oct 14;130(16):e140-2. doi: 10.1161/CIRCULATIONAHA.113.005819. No abstract available. PMID 25311622
- [Background] Spanos K, Tsilimparis N, Kolbel T. Exercise after Aortic Dissection: to Run or Not to Run. Eur J Vasc Endovasc Surg. 2018 Jun;55(6):755-756. doi: 10.1016/j.ejvs.2018.03.009. Epub 2018 Mar 31. No abstract available. PMID 29615314
- [Background] Boodhwani M, Andelfinger G, Leipsic J, Lindsay T, McMurtry MS, Therrien J, Siu SC; Canadian Cardiovascular Society. Canadian Cardiovascular Society position statement on the management of thoracic aortic disease. Can J Cardiol. 2014 Jun;30(6):577-89. doi: 10.1016/j.cjca.2014.02.018. Epub 2014 Feb 28. PMID 24882528
- [Background] Chaddha A, Kline-Rogers E, Braverman AC, Erickson SR, Jackson EA, Franklin BA, Woznicki EM, Jabara JT, Montgomery DG, Eagle KA. Survivors of Aortic Dissection: Activity, Mental Health, and Sexual Function. Clin Cardiol. 2015 Nov;38(11):652-9. doi: 10.1002/clc.22418. PMID 26769699
- [Background] Ghadieh AS, Saab B. Evidence for exercise training in the management of hypertension in adults. Can Fam Physician. 2015 Mar;61(3):233-9. PMID 25927108
- [Background] Li J, Boyd A, Huang M, Berookhim J, Prakash SK. Safety of exercise for adults with thoracic aortic aneurysms and dissections. Front Sports Act Living. 2022 Aug 22;4:888534. doi: 10.3389/fspor.2022.888534. eCollection 2022. PMID 36072558
- [Background] Meinlschmidt G, Berdajs D, Moser-Starck R, Frick A, Gross S, Schurr U, Eckstein FS, Hunziker S, Schaefert R. Perceived Need for Psychosocial Support After Aortic Dissection: Cross-Sectional Survey. J Particip Med. 2020 Jul 6;12(3):e15447. doi: 10.2196/15447. PMID 33064108
- [Background] Hays RD, Spritzer KL, Schalet BD, Cella D. PROMIS(R)-29 v2.0 profile physical and mental health summary scores. Qual Life Res. 2018 Jul;27(7):1885-1891. doi: 10.1007/s11136-018-1842-3. Epub 2018 Mar 22. PMID 29569016
- [Background] Eston RG, Davies BL, Williams JG. Use of perceived effort ratings to control exercise intensity in young healthy adults. Eur J Appl Physiol Occup Physiol. 1987;56(2):222-4. doi: 10.1007/BF00640648. PMID 3569229